CLINICAL TRIAL: NCT05759910
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Study of the Effect of BrainPhyt High Dose on Cognitive Function in Healthy Older Individuals
Brief Title: Effect of BrainPhyt High Dose on Cognitive Function in Healthy Older Individuals
Acronym: PHAEO-FOUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microphyt (Industry)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB2021-1360F
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Age-associated Memory Impairment
Keywords: Elderly; Microalgae; Cognitive function; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 4 capsules per day containing 275mg of Maltodextrin
  Interventions: Dietary Supplement: Placebo
- BrainPhyt High dose (Experimental): 4 capsules per day containing 275mg of BrainPhyt
  Interventions: Dietary Supplement: Brainphyt high dose

INTERVENTIONS:
Dietary Supplement: Brainphyt high dose — Participants will take BrainPhyt capsules during 3 months
  Arms: BrainPhyt High dose
Dietary Supplement: Placebo — Participants will take placebo capsules during 3 months
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate if BrainPhyt, a microalgae based ingredient may affect cognitive function parameters in older healthy individuals with evidence of age-related cognitive decline.

In a double blind, randomized manner, 40 free living males and females between 55 to 75 years with age-associated memory decline will ingest Brainphyt supplement or Placebo for 12 weeks. Cognitive function battery will be realized after 4 and 12 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent and to consume the investigational product daily for the duration of the study.
* Healthy males and females aged ≥ 55 and ≤ 75 years old.
* Body-mass index between 18.5 and 35.0 kg/m2
* Is free-living (living in a private home, alone or with family, and able to maintain their health and hygiene without assistance).
* Have age-associated memory impairment (AAMI) based on the following National Institute of Mental Health criteria, specified as scoring:

  1. Absence of dementia as determined by a score of >24 on the Mini Mental State Examination (MMSE).
  2. ≤29 or ≤9 on the VPA I and II portions of the Wechsler Memory Scale IV, respectively
  3. A score on the MAC-Q of ≥25.
* Is in general good health, as determined by the investigator
* Ability to comply and understand the cognitive function practice tests
* Willing to maintain their habitual diet and exercise routines.
* Willing to maintain consistent sleep duration the evening before study visits.

Exclusion Criteria:

* Use of medications or supplements known to alter cognitive function within past 2 weeks
* Abnormal clinical laboratory test that may affect study outcome.
* History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, gastrointestinal, pancreatic, or neurological disorders (including sleep disorders, head injuries, Alzheimer's disease, Parkinson's disease, stroke, inflammatory brain disease
* History or presence of cancer, except nonmelanoma skin cancer
* Uncontrolled hypertension/diabetes
* History of depression within past 24 months or use of psychotropic medications within 1 month of screening
* Planned major changes in lifestyle (i.e. diet, dieting, exercise level, travelling) during the duration of the study.
* History within previous 12 months of alcohol or substance abuse.
* History of heavy smoking (>1 pack/day) within past 3 months

Ages: 55 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in spatial Working Memory | From week 0 to week 12
  Mean Span Score in Corsi Blocks module of the COMPASS

SECONDARY OUTCOMES:
Change in spatial working memory | From week 0 to week 4
  Mean Span Score in Corsi Blocks module of the COMPASS
Change in attention and vigilance | From week 0 to week 12
  Mean reaction time and accuracy in Digit Vigilance Task module of the COMPASS
Change in attention and vigilance | From week 0 to week 4
  Mean reaction time and accuracy in Digit Vigilance Task module of the COMPASS
Change in executive function | From week 0 to week 12
  Mean reaction time and accuracy in Stroop task module of the COMPASS
Change in executive function | From week 0 to week 4
  Mean reaction time and accuracy in Stroop task module of the COMPASS
Change in episodic memory | From week 0 to week 12
  Mean reaction time and accuracy in Stroop task module of the COMPASS
Change in episodic memory | From week 0 to week 4
  Mean reaction time and accuracy in Stroop task module of the COMPASS
Change in perceptual and cognitive skills | From week 0 to week 4
  Mean reaction time and accuracy in Neurotracker light reaction test
Change in perceptual and cognitive skills | From week 0 to week 12
  Mean reaction time and accuracy in Neurotracker light reaction test
Stress level | From week 0 to week 4
  Change in Cohen's Perceived Stress Scale from 0 to 40 (high stress)
Stress level | From week 0 to week 12
  Change in Cohen's Perceived Stress Scale from 0 to 40 (high stress)
Sleep quality | From week 0 to week 12
  Change in Leeds Sleep Evaluation questionnaire from 0 to 10 (low sleep quality)
Sleep quality | From week 0 to week 4
  Change in Leeds Sleep Evaluation questionnaire from 0 to 10 (low sleep quality)
Mood state | From week 0 to week 4
  Change Bond-Lader Mood rating scale from 0 to 10 (low mood state)
Mood state | From week 0 to week 12
  Change Bond-Lader Mood rating scale from 0 to 10 (low mood state)
Inflammation IL-6 | from week 0 to week 12
  Change Interleukin-6 level (pg/ml)
Inflammation IL-6 | from week 0 to week 4
  Change Interleukin-6 level (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoo C, Maury J, Gonzalez DE, Ko J, Xing D, Jenkins V, Dickerson B, Leonard M, Estes L, Johnson S, Chun J, Broeckel J, Pradelles R, Sowinski R, Rasmussen CJ, Kreider RB. Effects of Supplementation with a Microalgae Extract from Phaeodactylum tricornutum Containing Fucoxanthin on Cognition and Markers of Health in Older Individuals with Perceptions of Cognitive Decline. Nutrients. 2024 Sep 5;16(17):2999. doi: 10.3390/nu16172999. PMID 39275314